CLINICAL TRIAL: NCT04664725
Title: A Single-center, Open-label, Fixed-sequence Phase I Drug-drug Interaction Clinical Study to Investigate the Pharmacokinetics of SHR3680 With Repaglinide (CYP2C8 Substrates) and Bupropion (CYP2B6 Substrates) in Prostate Cancer Patients
Brief Title: Drug-drug Interaction of SHR3680 With Repaglinide and Bupropion
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SHR3680-I-DDI-02
Record Dates: First submitted 2020-11-22; First posted 2020-12-11 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-11

CONDITIONS: Prostate Cancer Patients
MeSH Terms: interventions — repaglinide; Bupropion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR3680+ Repaglinide, Bupropion (Experimental): * Experimental: Repaglinide, Bupropion and SHR3680
  * Repaglinide and Bupropion QD on Day 1 and Day 21, SHR3680 240 mg once daily (QD) from Study Day 6 - 26
  Interventions: Drug: Repaglinide, Bupropion and SHR3680

INTERVENTIONS:
Drug: Repaglinide, Bupropion and SHR3680 — Single dose of oral administration of Repaglinide and Bupropion, Multiple dose of oral of SHR3680

SUMMARY:
The DDI study had been designed to investigate the effect of SHR3680 on the pharmacokinetics of Repaglinide and Bupropion

ELIGIBILITY:
Inclusion Criteria:

* 1. 18 ≤ age ≤75, male;
* ECOG score of physical condition is 0 ~ 1;
* The expected survival time is at least 3 months;
* Prostatic adenocarcinoma confirmed by histological or cytological examination, with no indication of neuroendocrine or small-cell characteristics;
* Fasting blood glucose level is: 3.9～6.1mmol/L；
* The functional level of organs must meet the following requirements (no blood transfusion or hematopoietic growth factor treatment was received within 2 weeks before routine blood screening) :

  * ANC ≧ 1.5 x 109 / L;
  * PLT ≧ 80 x 109 / L;
  * Hb ≧ 90 g/L;
  * TBIL ≦1.5 x ULN;
  * ALT and AST≦2.5×ULN;
  * BUN and Cr ≦1.5 x ULN;
  * GFR ≧ 60 ml/min / 1.73 m2.
* According to the researcher's judgment, it can comply with the experimental scheme;
* Volunteer to participate in this clinical trial, understand the study procedures and have signed informed consent.

Exclusion Criteria:

* Any previous anti-tumor therapy (including radiotherapy, chemotherapy, surgery, molecular targeted therapy, immunotherapy, etc.), except ADT therapy, shall be completed until the washout period of the first drug administration in this study is <4 weeks;
* Plan to receive any other anti-tumor therapy during the study;
* As subjects, to participate in other drug clinical trials, the last trial drug administration is less than 4 weeks from the first administration of the drug in this study;
* The presence of intracerebral tumor lesions according to imaging diagnosis;
* Have a history of epilepsy, or have diseases that can induce epileptic seizures within 12 months before the first administration of the drug in this study (including a history of transient ischemic attack, cerebral stroke (except cerebral ischemia lesions found by simple imaging examination), and need to be hospitalized with cerebral trauma and consciousness disorder);
* Active heart disease, including severe/unstable angina, myocardial infarction, symptomatic congestive heart failure, and drug-requiring ventricular arrhythmias, within 6 months prior to the first administration of the drug in this study;
* Inability to swallow, chronic diarrhea and ileus, history of gastrointestinal surgery, or other factors affecting drug use and absorption as determined by the investigator;
* Patients with active HBV or HCV infection (HBV copy count ≥ 104 copies /mL, HCV copy count ≥ 103 copies /mL) and active syphilis;
* A history of immunodeficiency (including HIV positive, other acquired or congenital immunodeficiency diseases) or a history of organ transplantation;
* Patients who were unwilling to use effective contraceptive methods during the whole study treatment period and within 3 months after the last administration;
* Allergic constitution, including a history of severe drug allergy or drug allergy;
* Screening for excessive smoking in the first 6 months (≥5 cigarettes/day) or smoking within 48 hours before the first dose, or not interrupting smokers during the main study trial, and screening for drug use in the first 3 months with a history of drug abuse or positive drug abuse screening;
* has a history of alcoholism or within 6 months prior to screening often drinkers, namely the essence of drinking more than 14 units of alcohol a week (1 = 360 mL of alcohol content of 5% beer or 45 mL of 40% alcohol liquor or 150 mL wine alcohol content of 12%) or within 48 h before taking the medicine for the first time drinking, or D - 1 in the alcohol breath test positive, or the body can't stop alcohol intake during the study period;
* Use of any vitamin product, health product or herb 14 days prior to the first administration;
* Ingestion of grapefruit or fruit juice products such as grapefruit, foods or beverages containing caffeine, xanthine or alcohol within 48 hours before taking the study drug;Strenuous exercise, or other factors affecting drug absorption, distribution, metabolism, and excretion;
* Within 2 weeks before the first drug uptake, uptake CYP2C8 and CYP2B6 inhibitors were used, or drugs affecting gastric acid secretion.;
* abnormal coagulation function at screening stage (INR >1.5 or prothrombin time (PT) > ULN+4 seconds or APTT> 1.5uln), bleeding tendency or thrombolytic therapy;
* Repaglinide contraindications (insulin-dependent -IDDM, C-peptide-negative diabetic patients, diabetic ketoacidosis with or without coma);
* Contraindications to bulimia or anorexia (epileptic history, bulimia or anorexia, abstinence from alcohol or sedatives suddenly);
* Those with a history of fainting needle or blood, have difficulty in blood collection or cannot tolerate vein puncture for blood collection;
* Concomitant diseases (such as poorly controlled hypertension, severe diabetes, thyroid disease, psychosis, etc.) or any other conditions that, in the investigator's judgment, would seriously endanger the patient's safety or affect the patient's completion of the study.

Ages: 45 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Peak Plasma Concentration(Cmax) | Day1 and Day21
  Summary of Pharmacokinetic parameters Maximum Plasma concentration (Cmax) for Repaglinide and Bupropion
Area under the plasma concentration versus time curve(AUC0-t) | Day1 and Day21
  Summary of Pharmacokinetic parameters Area Under the Plasma Concentration-time Curve form 0 to any time before the last quantifiable concentration(AUC0-t)for Repaglinide and Bupropion

CONTACTS AND LOCATIONS:
Overall Officials: Weiqing Han, Ph.D, Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dai T, Xu Z, Huang L, Wang Y, Zeng G, Ye M, Liu K, Zeng F, Jiang S, Han W, Cao J. A single-centre, open-label, single-arm, fixed-sequence pharmacokinetic study of SHR3680 on repaglinide and bupropion in prostate cancer patients. Br J Clin Pharmacol. 2023 Feb;89(2):874-886. doi: 10.1111/bcp.15528. Epub 2022 Oct 9. PMID 36098470